CLINICAL TRIAL: NCT06343753
Title: Quality of Recovery After Laparoscopic Cholecystectomy: A Prospective, Randomised, Controlled Trial Comparing Opioid Free Multimodal Analgesia Versus Opioid Based Anesthesia
Brief Title: Quality of Recovery After Laparoscopic Cholecystectomy Comparing Opioid Free Analgesia Versus Opioid Free Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Samy, Doctor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: FMASU MD46/2024
Record Dates: First submitted 2024-03-19; First posted 2024-04-03 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Quality of Recovery; Pain, Postoperative; Elective Laparoscopic Cholecystectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine; Lidocaine; Ketamine; Bupivacaine; Ondansetron; Metoclopramide; Propofol; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opioid free anesthesia (OFA) group (Active Comparator): Analgesia will be provided by syringe containing ketamine, Lidocaine and Dexmedetomidine in induction and maintenance according to lean body weight (LBW).
  Induction :
  Ketamine: 0.5 mg/kg (IBW), Lidocaine 1 mg/kg and dexmedetomidine 0.5 mg/kg (LBW) for induction to be given in 10 ml syringe over 10 minutes.
  Maintenance : The maintenance mixture" - 50 cc syringe containing:
  50 mcg Dexmedetomidine (0.5 cc of standard 100 mcg/ml solution) 50 mg Ketamine 500 mg Lidocaine (25 ml of standard 2% solution) NaCl up to total 50 ml
  Interventions: Drug: Opioid free analgesia
- Opioid based anesthesia( OBA )group (Active Comparator): Fentanyl 2 g/kg (LBW) as induction dose in 10 ml syringe to be given over 10 minutes, and 1 g/kg/h in 50 ml syringe as infusion during operation starting before skin incision for Group TBA.
  Interventions: Drug: Opioid based Anesthesia

INTERVENTIONS:
Drug: Opioid free analgesia — o Group OFA: Opioid free anesthesia Analgesia will be provided by syringe containing ketamine, Lidocaine and Dexmedetomidine in induction and maintenance according to lean body weight (LBW).
  Other Names: Dexmedetomidine; Lidocaine; Ketamine; Bupivacaine; Ondansetron; Metoclopramide; Propofol
  Arms: Opioid free anesthesia (OFA) group
Drug: Opioid based Anesthesia — o Group TBA: Traditional balanced anesthesia Analgesia will be provided by fentanyl in induction and maintenance according to Ideal Body Weight (IBW)
  Other Names: Fentanyl; Propofol; Ondansetron; Metoclopramide; Bupivacaine
  Arms: Opioid based anesthesia( OBA )group

SUMMARY:
The aim of this study is to compare the quality of recovery from general anesthesia and surgery using the quality of recovery 15 item scale (QoR-15) for participant's receiving opioid-Sparing anesthesia with those receiving standard opioid-containing anesthesia in Patients undergoing a scheduled laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Type of Study: interventional, randomized and double-blinded controlled trial. Study Setting: The operating theatres of Ain Shams University Hospitals. Study Period: over one year.

Study Procedures

Patients will be randomly allocated by computer generated randomization and using opaque sealed envelopes to one of the two groups according to the used analgesia into:

o Group Traditional balanced anesthesia (TBA): Analgesia will be provided by fentanyl in induction and maintenance according to Ideal Body Weight (IBW)

o Group Opioid free anesthesia (OFA): Analgesia will be provided by syringe containing ketamine, Lidocaine and Dexmedetomidine in induction and maintenance according to lean body weight (LBW).

Both groups will receive port site infiltration with bupivacaine 0.25% 20 ml.

Pre-operatively, all patients will receive Ondansetron 4 mg IV, and metoclopramide 10 mg intravenously (IV).

After proper assessment of the airway and anticipation of difficult airway, all patients will receive midazolam 2 mg IV for sedation and we will start pre-oxygenation with 100% O2 on 8 L/min for 3 min via face mask.

All patients will receive general anesthesia induction by propofol 1.5-2 mg/kg (LBW), analgesia according to patient group, and muscle relaxation by atracurium 0.5 mg/Kg LBW to facilitate endotracheal intubation. Anesthesia will be maintained by isoflurane whose concentration will be adjusted according to patient's hemodynamics. Analgesia used in the study will be prepared in the pharmacy and will be given a code so that the anesthetist in charge will be blinded to the randomisation group and the analgesia used. The analgesia will be prepared as follows:

* Fentanyl 2 mg/kg (LBW) as induction dose in 10 ml syringe to be given over 10 minutes, and 1 mg/kg/h in 50 ml syringe as infusion during operation starting before skin incision for Group TBA.
* Group OFA :

Induction :

Ketamine: 0.5 mg/kg (IBW), Lidocaine 1 mg/kg and dexmedetomidine 0.5 mg/kg (LBW) for induction to be given in 10 ml syringe over 10 minutes.

Maintenance : The maintenance mixture" - 50 cc syringe containing:

50 mcg Dexmedetomidine (0.5 cc of standard 100 mcg/ml solution) 50 mg Ketamine 500 mg Lidocaine (25 ml of standard 2% solution) NaCl up to total 50 ml. Ketamine 0.1 mg/kg/h (IBW), Lidocaine 1 mg/kg/h and dexmedetomidine 0.1 mg/kg/h (LBW) as infusion during operation starting before skin incision. (1ml/10 kg of solution from "The maintenance mixture" syringe ) After skin preparation and before port insertion, 20 ml of 0.25% bupivacaine solution was infiltrated through the abdominal wall 4ml around each port site in both groups.

About 15 min before the end of the operation reduce maintenance dose to 0.5 ml/10 kg/h Ventilator Settings: the ventilation will be achieved with a volume-controlled mode ventilation, respiratory rate adjusted according to EtCO2 to range between 35-45 mmHg, a tidal volume of 6-8 ml/kg and mixture of gases in proportion 50% oxygen and 50% air, with PEEP 5 cm H2O using a closed circle system and with a total fresh gas flow rate of 3L/min.

Analgesic infusion will be stopped after skin closure. Paracetamol 1 gm and diclofenac 75 mg (incorporated in IV infusion fluids) will be given intra-operatively before emergence.

At the end of surgery, muscle relaxation will be reversed with neostigmine (up to 5 mg) and atropine (up to 2 mg).

These procedures will be done by supervisors and experts. Patients will be kept after extubation for observation in PACU until fulfilling an Aldrete score of 9.

Patients will receive metoclopramide 10 mg intravenously (IV) and Ondansetron 4 mg IV as post-operative nausea and vomiting (PONV) treatment.

Post-operative analgesia will be offered in regular doses of paracetamol 1 gm IV every 6 hours for the following 24 hours, and rescue doses of IV nalbuphine 5 mg (Up to 20 mg max/dose). If VAS score is >3.

The anesthetist evaluating outcomes in PACU and in the ward will not participate in the anesthesia and will not be aware of the randomisation group.

ELIGIBILITY:
Inclusion criteria :

* Age group: 18-65 year of both sex.
* Patients with ASA (American society of anesthesiologist) classification I-II.
* Undergoing a scheduled laparoscopic cholecystectomy

Exclusion Criteria:

* Pregnant or breast-feeding women
* ASA physical status class > 2
* The need to change laparoscopic surgery to an open one
* Allergy to any of the drugs used in the study
* local skin infection at the trocar injection site
* 1st or 2nd degree Heart block
* Chronic treatment by beta-blockers
* HR <50 bpm
* Epilepsy or seizures
* Alcohol or drug abuse
* Psychiatric disease
* History of chronic pain

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-09-20 (Actual)

PRIMARY OUTCOMES:
Quality of recovery | 24 hour
  The 15-item quality of recovery (QoR-15) score at 24 h postoperatively.
  o The QoR-15 score : is a shorter validated version of the QoR-40 and provides an efficient evaluation of post-operative recovery from the participant's perspective with total QoR-15 score ranging from 0 (extremely poor recovery) to 150 (excellent recovery).(Stark et al.,2013) Each question is measured on a Likert scale ranging from 0-10; where 0 = none of the time [poor] to 10 = all of the time [excellent]. Results are considered clinically significant if there is a change of score of eight.

SECONDARY OUTCOMES:
Post operative pain | 24 hour
  Postoperative pain score for 24 hours using the Visual Analogue Scale (VAS): 30 min after recovery, hourly for 2 h and every 6 h for 24 h.
  The Visual Analogue Scale (VAS) consists of a 10 cm straight line with the endpoints defining extreme limits of 'no pain at all' (0 cm) and 'pain as bad as it could be' (10 cm). The patient is asked to mark his pain.
  Level on the line between the two endpoints. The distance between 0 and the mark then defines the subject's pain score. A higher score indicates greater pain intensity.
  Nalbuphine consumption during the 24 hours following extubation.
Postoperative Hypoxia | 24 hour
  Number of patients who will experience The occurrence of a severe postoperative opioid-related adverse event within the first 24 hours after extubation such as:
  Postoperative hypoxemia defined as peripheral oxygen saturation (SpO2) <92% on room air with a need for oxygen supplementation; the duration of oxygen treatment will be also recorded.
Postoperative nausea and vomiting | 24 hour
  Number of patients sustains episodes of PONV.
Postoperative bradycardia | 24 hour
  Number of patients sustains Bradycardia (defined as: HR ≤50 bpm), atropine 0.6 mg/kg increments will be administered till acceptable response.
Postoperative hypotension | 24 hour
  Number of patients sustains Hypotension (defined as a decrease in systolic blood pressure >20% of baseline value), administration of ephedrine5-6 mg increments, 250 ml fluid bolus IV and reduction of analgesic maintenance infusion by 50% will be initiated till acceptable response.
Postoperative hypertension | 24 hour
  Number of patients sustainsHypertension (defined as an increase in systolic blood pressure >20% of baseline value),bolus of the analgesic maintenance infusion then elevation of the infusion rate by 50% will be administered till acceptable response after exclusion of causes other than sympathetic response to surgical stimulus .

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No